CLINICAL TRIAL: NCT07018791
Title: Assessment of the Impact of Art-Based Pain Assessment Tool on Pain Communication, Joint Function, and Anxiety in Patients With Temporomandibular Joint Disorders: A Randomized Controlled Trial
Brief Title: Art-Based Pain Assessment Tool in Patients With Temporomandibular Joint Disorders
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Razan Baabdullah, Assistant professor of oral and maxillofacial surgery, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 02-01-25
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Temporomandibular Disorders (TMD); Wilkes 1 and 2; TMJ Pain; TMJ - Oral &Amp;Maxillofacial Surgery; Art Therapy; TMD Art Pain Study
Keywords: Temporomandibular joint disorders; Artistic Pain Exploration (APE); Visual Pain Expression; Art-Based Assessment; Multisensory Pain Assessment; Randomized Controlled Trial; Pain Communication; Patient-Reported Outcomes; TMJ Function
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Individuals analyzing the results (comparing scores on pain communication, anxiety, and TMJ pain and function) are blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in this group receive standard care for Temporomandibular Joint Disorders (TMD), which includes a clinical examination, assessment of pain using the Visual Analogue Scale (VAS), anxiety and depression screening (GAD-7 and PHQ-9), evaluation of jaw pain and function, and conservative treatment through medication and self-care instructions.
  Interventions: Diagnostic Test: Standard TMD Assessment
- Intervention Group (Experimental): Participants in this group receive the same standard care as the control group, with the addition of an art-based method designed to enhance the understanding and communication of pain.
  Interventions: Diagnostic Test: Standard TMD Assessment; Diagnostic Test: Artistic Pain Exploration (APE) Method

INTERVENTIONS:
Diagnostic Test: Standard TMD Assessment — This is the conventional diagnostic and management approach for TMD, focusing on physical evaluation and symptom tracking without the use of any visual or art-based tools. It serves as the baseline for comparison in this study.
Diagnostic Test: Artistic Pain Exploration (APE) Method — This approach involves showing patients three expressive paintings and asking them to select the one that best resonates with them. A guided interview follows, using the artwork to explore the patient's pain characteristics, emotional impact, and functional limitations. This method aims to provide a richer, more personalized understanding of the patient's pain experience.
  Other Names: Art-based assessment tool
  Arms: Intervention Group

SUMMARY:
Title of Study:

Assessment of the Impact of Art-Based Pain Assessment Tool on Pain Communication, Joint Function, and Anxiety in Patients with Temporomandibular Disorders (TMD): A Randomized Controlled Trial

Location:

King Abdulaziz University Dental Hospital (KAUFD), Jeddah, Saudi Arabia What Is This Study About?

This study examines how an art-based tool can help improve communication and understanding of pain among patients with jaw joint disorders (TMD). It compares two groups:

* Standard care: Routine diagnostic and therapeutic procedures
* Intervention: Standard care plus a guided art-based tool using paintings to express and discuss the TMD experiences What Is the Art-Based Tool?

This novel method, called the Artistic Pain Exploration (APE), uses paintings to help patients describe their pain that relates to TMD and its effect on their quality of life:

1. Participants will be shown three paintings (e.g., The Scream by Edvard Munch)
2. Participants will choose the one that best resonates with them
3. A guided discussion follows, exploring how the image relates to their physical and emotional pain as well as the effect of pain on their daily activities

Research Questions:

1. Does using the APE method help participants better communicate and understand their pain?
2. Does it improve jaw function and reduce anxiety more than standard assessment? Who Can Participate?

Participants may be eligible if they:

* Are 18 years or older
* Have early-stage TMD (not needing surgery)
* Can give informed consent

Participants cannot participate if they:

* Require jaw surgery
* Have severe mental illness (e.g., psychosis or bipolar disorder)
* Take narcotic pain medications regularly What Will Happen During the Study?
* Participants are randomly assigned to one of the two groups.
* Each participant will complete a standardized questionnaire before and after two weeks to assess the level of anxiety.
* All participants will be screened for depression via a standardized questionnaire before the first visit.
* All will undergo a clinical exam to assess the TMJ pain and function and receive appropriate medications and lifestyle instructions.
* Some participants (intervention group) will also discuss their pain using the artwork.
* All participants will be seen for a follow up in 2 weeks to assess the TMJ function and pain.

Potential Risks and Discomforts

Participants may experience:

* Emotional discomfort while discussing pain
* Mild anxiety during interviews or questionnaires If needed, a psychiatrist on the research team will provide support or referrals.

Potential Benefits

* A better understanding of pain
* Improved communication with care provider
* Possible improvement in pain and jaw function

Costs There are no costs to participate. All treatments are provided free of charge.

Compensation / Treatment for Injury

* If participants experience harm from this study, necessary medical care will be provided by the research team.
* No financial compensation will be provided by King Abdulaziz University.

Confidentiality Participants' identity and medical records will remain confidential. Only approved researchers and auditors will have access to data, in accordance with applicable laws. Any results published will not include participants' name or identifying details.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Diagnosed with Temporomandibular Disorders (TMD) requiring conservative management only and classified as Wilkes' stage I or II
* Able to understand and sign the informed consent form

Exclusion Criteria:

* Patients requiring surgical intervention for TMD
* Presence of severe mental illness, such as psychotic disorders or bipolar affective disorders
* Regular use of narcotic (opioid) pain medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Patient-reported outcomes on pain understanding and communication | Baseline
  The Pain Communication and Understanding Questionnaire is a validated tool designed to assess how well patients understand their own pain and how effectively they are able to communicate that experience with their healthcare provider.

SECONDARY OUTCOMES:
Pain Level | At baseline and 2-week follow-up.
  Measured by the Visual Analogue Scale (VAS), this outcome captures the intensity of pain as reported by the patient on a scale from 0 (no pain) to 10 (worst pain imaginable).
Temporomandibular Joint (TMJ) Function | At baseline and 2-week follow-up.
  TMJ functional capacity will be evaluated through a set of clinical assessments:
  Maximal interincisal distance (mm): measured as the maximum unassisted vertical opening between the incisal edges of upper and lower central incisors using a calibrated ruler or caliper.
  Mandibular excursive and protrusive movements (mm): lateral and anterior movements will be measured from centric occlusion to maximum displacement.
  Pain on mouth opening (VAS 0-10): Participants will rate pain intensity during maximum mouth opening using a 10-point visual analog scale.
  Presence of joint sounds (clicking/crepitus): assessed through bilateral palpation and auscultation during mandibular motion; recorded as Present or Absent.
  Presence of occlusal wear facets: identified through intraoral examination; recorded as Present or Absent.
  Muscle of mastication tenderness: evaluated via bilateral palpation of the muscles of mastication and recorded as tender or non-tender.
Anxiety level | At baseline and 2-week follow-up
  Assessed using the General Anxiety Disorder-7 (GAD-7) questionnaire, this outcome indicates the severity of anxiety symptoms experienced by the patient. The minimum score is zero and the maximum is 21. Lower scores mean lower anxiety levels.
Depression Screening | At baseline only.
  Screened at baseline using the Patient Health Questionnaire-9 (PHQ-9), this outcome identifies the presence and severity of depressive symptoms in the patient. The minimum score is zero and the maximum is 27. Lower PHQ-9 scores indicate fewer or less severe depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University, Faculty of Dentistry, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Al-Khotani A, Naimi-Akbar A, Gjelset M, Albadawi E, Bello L, Hedenberg-Magnusson B, Christidis N. The associations between psychosocial aspects and TMD-pain related aspects in children and adolescents. J Headache Pain. 2016;17:30. doi: 10.1186/s10194-016-0622-0. Epub 2016 Apr 5. PMID 27044436
- [Result] Wilson C, Bungay H, Munn-Giddings C, Boyce M. Healthcare professionals' perceptions of the value and impact of the arts in healthcare settings: A critical review of the literature. Int J Nurs Stud. 2016 Apr;56:90-101. doi: 10.1016/j.ijnurstu.2015.11.003. Epub 2015 Nov 27. PMID 26696399
- [Result] Regev D, Cohen-Yatziv L. Effectiveness of Art Therapy With Adult Clients in 2018-What Progress Has Been Made? Front Psychol. 2018 Aug 29;9:1531. doi: 10.3389/fpsyg.2018.01531. eCollection 2018. PMID 30210388
- [Result] Kirkham JA, Smith JA, Havsteen-Franklin D. Painting pain: an interpretative phenomenological analysis of representations of living with chronic pain. Health Psychol. 2015 Apr;34(4):398-406. doi: 10.1037/hea0000139. PMID 25822055

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT07018791/Prot_SAP_000.pdf